CLINICAL TRIAL: NCT03398486
Title: Evaluation of the Effectiveness of Kinesiotaping and Inactivation of Trigger Points in Chronic Myofascial Pain of Temporomandibular Joint Dysfunction
Brief Title: The Effectiveness of Kinesiotaping and Inactivation of Trigger Points in Chronic Myofascial Pain of TMD
Acronym: KT/TrP/TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Ministry of Health, Poland (Other Government)
Responsible Party: Principal Investigator, Edward Kijak, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-0012/36/15
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Myofascial Pain; TMD
Keywords: Kinesiotaping, Manual therapy; Physiotherapy

STUDY DESIGN:
Intervention Model Description: 1. Experimental: Kinesiotaping Participants receive an application of active tapes (KT) Original kinesiotaping active tapes Duration: 2 times Application maintenance 5 days with a break for the weekend Muscle application on the masseter muscle area, using a tape (5 cm wide) dissected into 2 parts called tails, which included the treatment site without their tension.
  Experimental: active inactivation of trigger points (TrP) Duration: 10-20 minutes of surgery; 2 inactivation treatments Between the treatments 5 days break
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping (Experimental): Original kinesiotaping active tapes Duration: 2 times Application maintenance 5 days with a break for the weekend Muscle application on the masseter muscle area, using a tape (5 cm wide) dissected into 2 parts called tails, which included the treatment site without their tension.
  Interventions: Diagnostic Test: Kinesiotaping
- inactivation of trigger points (TrP) (Experimental): Duration: 10-20 minutes of surgery; 2 inactivation treatments Between the treatments 5 days break
  Interventions: Diagnostic Test: inactivation of trigger points (TrP)

INTERVENTIONS:
Diagnostic Test: Kinesiotaping — Dynamic adhesive taping is a method that involves the application of specific tapes to the surface of the patient's skin in order to use the natural self-healing processes of the body. It is often used as an element that sustains the therapeutic effect. Its action is based mainly on the action normalizing muscle tone, supporting the work of joints, improving the function of weakened muscles, increasing microcirculation at the site of application.
  Other Names: Dynamic adhesive plaster, Dynamic adhesive tape
  Arms: Kinesiotaping
Diagnostic Test: inactivation of trigger points (TrP) — A procedure for releasing trigger points using physiotherapy using the ischemic compression method, which involves applying pressure to the active trigger point, until it is switched off, i.e. pain ceases.The location of the trigger point is done palpatively, with a pliers grip, covering the strained tissue on the inside and outside of the cheek with the thumb and index finger.
  Other Names: compressive mobilization
  Arms: inactivation of trigger points (TrP)

SUMMARY:
In patients with a long-lasting TMD syndrome, especially of a muscular nature, palpation examination can locate the trigger points of pain (TrP) in the chewing muscles, i.e., the nodules in the shape of bumps the size of rice or pea grains. Kinesiotaping (KT) is considered as an intervention method that can be used to release latent myofascial trigger points. It is a method that involves applying specific tapes to the patient's skin surface in order to use the natural self-healing processes of the body. The aim of the study was to evaluate the effect of Kinesiotaping methods and inactivation of Trigger Points on nonpharmacological elimination of pain in patients with functional disorders of the masticatory motor system.

DETAILED DESCRIPTION:
BACKGROUND:

Temporomandibular Dysfunction (TMD) is a disease characterized by a set of signs and symptoms that may include joint noise, pain in the mastication muscles, limitation of mandibular movements, facial pain, joint pain and / or dental wear. Pain appears as a very present and striking symptom, with a tendency to chronicity. This is a difficult treatment condition often associated with psychological factors such as anxiety. In patients with a longlasting TMD syndrome, especially those of a muscular nature, palpation can locate the trigger points of pain (TrP) in the chewing muscles, i.e. the nodules in the shape of bumps the size of grains of rice or peas. Of particular importance in the treatment of pain syndromes of temporomandibular joint disorders is physiotherapy and physical therapy. Some studies have shown improvement in subjects with chronic pain using different physiotherapy treatments, but this requires further investigation to determine the effectiveness of individual therapies in the fight against pain.

PROBLEM:

The multiple manifestation of symptoms causes a multitude of treatment methods and indicates that there is still no consensus in the understanding of the pathophysiology of the underlying TMD mechanisms. Treatment of pain syndrome in temporomandibular dysfunction due to heterogeneity of causes should have a multiprofile character. Despite the wide range of strategies used to treat patients with TMD, some patients have a temporary and / or unsatisfactory relief response. There are many physiotherapeutic methods to fight pain, among others: compressive mobilization, positional release, myofascial relaxation, active relaxation technique, postisometric relaxation technique. Of the commonly used methods, a deep tissue massage and stretching. Some of them are very unpleasant for patients, because in the first phase they intensify pain, eg active inactivation (therapy) of trigger points (TrP). Kinesiotaping is a painless method that does not intensify pain symptoms. Reports from various researchers are contradictory in this regard, hence the attempt to compare both methods in the aspect of non-pharmacological analgesic activity in patients with TMD.

HYPOTHESIS:

Researchers believe that in patients with severe pain symptoms, patients with TMD who are often accompanied by anxiety before symptom intensification, it is very important to use physiotherapeutic methods, which can eliminate or reduce pain in a non-pharmacological manner. In this type of patients, the psychological aspect is important in the form of immediate relief without aggravating the symptoms at least in the first phase, because it can cause patients psychological reluctance to the entire treatment process. Because of the mutual influence between pain and psychological factors, it is expected that the analgesic effect will have a positive effect influence on the level of anxiety before further often long-term therapeutic treatment.

AIM:

Evaluation and comparison of the analgesic efficacy of two physiotherapeutic methods: Kinsiotapinng (KT) and active inactivation of trigger points (TrP) in the pain levels in individuals with chronic pain due muscular TMD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years, both male and female
* Provide informed consent to participate in the study;
* Having a diagnosis of muscular pain TMD(Temporomandibular Disorders) according to group -I A, axis I RDC/TMD(Research Diagnostic Criteria)
* Visual analogic scale (VAS) score from 4 to 10 for 14 days
* Not have history of alcohol or drugs abuse within the past 6 months as self-reported
* Not use ot carbamazepine (or similar) within the past 6 months as self reported
* Not have history of neurosurgery as self-reported
* Not have history of major psychiatric disorders such as schizophrenia and bipolar disorder
* Not have any other previously diagnosed disorder with symptoms similar to the TMD, such as fibromyalgia.

Exclusion Criteria:

* One absence during therapeutic sessions;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-02 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
1. Change from baseline in Visual Analogic Scale | 14 days
  The visual analogic scale allows us to convert subjective sensations as pain on numerical data. A 10cm scale where 0cm is no pain and 10cm the worse imaginable pain, will be used and the subjects will be asked to mark a point on the scale representing their pain. This instrument will be used to compare the VAS values before and after the intervention.

OTHER OUTCOMES:
1. Patient Global Impression of Change Scale (PGICS) | 3 months
  The Patient Global Impression of Change Scale (PGICS) is an understandable, adequate, easy-to-use instrument capable of measuring the perception of change in health status and satisfaction with the treatment of individuals with chronic musculoskeletal pain. It is a one-dimensional measurement instrument in which individuals rate their improvement associated with intervention on a 7-item scale ranging from 1 (no change) to 7 (Much better).

CONTACTS AND LOCATIONS:
Overall Officials: Edward S Kijak, DSc, Study Director — Pomeranian Medical University

IPD SHARING:
Plan to Share IPD: No